CLINICAL TRIAL: NCT01127477
Title: Examination of Volume Effect and Safety of 6 % Hydroxyethyl Starch 130/0.4 in Patients Undergoing Major Elective Surgery - an Uncontrolled, Open-labelled, Multi-centre Study
Brief Title: Study to Obtain Volume Effect and Safety Data on 6 % Hydroxyethyl Starch 130/0.4 in Pediatric and Adult Patients Undergoing Major Elective Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fresenius Kabi Japan (Industry)
Responsible Party: Sponsor
Organization: Fresenius Kabi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HE06-008-CP3
Record Dates: First submitted 2010-05-17; First posted 2010-05-21 (Estimated); Last update posted 2012-06-26 (Estimated); Status verified 2012-03

CONDITIONS: Plasma Volume Substitution (Hypovolemia) Including Massive Hemorrhage
Keywords: Hypovolemia, surgical blood loss
MeSH Terms: conditions — Hypovolemia; Blood Loss, Surgical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: 1: Hydroxyethyl starch 130/0.4, 6 %

INTERVENTIONS:
Drug: 1: Hydroxyethyl starch 130/0.4, 6 % — 1: Up to 50 ml 6 % hydroxyethyl starch 130/0.4/kg body weight administered intravenously from start of surgery (skin incision) until two hours after end of surgery.

SUMMARY:
The study shall evaluate the volume effect and safety of 6 % hydroxyethyl starch 130/0.4 for restoration and maintenance of hemodynamics during the investigational period in patients undergoing major elective surgery. Up to 50 mL 6% hydroxyethyl starch/kg body weight will be administered from start of surgery until two hours after end of surgery. The study hypothesis is that 6 % hydroxyethyl starch 130/0.4 will have a reliable volume effect and can be safely administered up to the dose limit.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing major elective surgery
* Adults patients (≥20 years of age): expected blood loss of ≥ 1000mL Pediatric patients (<20 years of age): expected blood loss ≥ 15 mL/kg
* Adult patients: Routine measurement of Central Venous Pressure (CVP)

Exclusion Criteria:

* Known or suspected allergy to hydroxyethyl starch, including its ingredients (inclusive corn) and related drugs
* ASA classification ≥ IV
* Adult patients: renal failure with oliguria (<400 mL urin /24hours) and anuria Pediatric patients: renal failure with oliguria and anuria not related to hypovolemia
* Known bleeding disorders
* Other contra-indications according to the current SmPC of Voluven 6% solution for infusion.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-05; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Volume Effect | Saved albumin: during surgery; Time course of hemodynamic stability: from end of surgery until 24 h after surgery
  Volume effect will be assessed by evaluating the following parameter:
  1. Saved albumin:
     For adult patients: Amount of 6 % hydroxyethyl starch 130/0.4 (HES130) administered during surgery once 1000 mL of HES130 are exceeded.
     For pediatric patients: Amount of HES130 administered during surgery once 10 mL HES130/kg body weight are exceeded.
  2. Time course of hemodynamic stability

SECONDARY OUTCOMES:
Fluid Balance | From one day before (pediatric patients)/ immediately before (adults) induction of anesthesia until 48 hours after end of surgery
  Fluid balance = fluid input vs. fluid output
Hemodynamics | From one day before (pediatric patients)/ immediately before (adults) induction of anesthesia until 48 hours after end of surgery
CVP | Immediately before or after induction of anesthesia (depending on routine procedures), every hour after skin incision, and 2 hours after surgery
  Central venous pressure (CVP); not mandatory for pediatric patients
Hematology | One day before (pediatric patients)/ immediately before (adults) induction of anesthesia, every hour after skin incision (adults), end of surgery (adults), 2 hours and 24 hours after end of surgery
Clinical Chemistry | One day before (pediatric patients)/ immediately before (adults) induction of anesthesia, end of surgery (adults), 2 hours after end of surgery (pediatric patients), and 24 hours after end of surgery
Hemostasis | One day before (pediatric patients)/ immediately before (adults) induction of anesthesia, end of surgery (adults), 2 hours and 24 hours after end of surgery
Body Temperature | One day before (pediatric patients)/ immediately before (adults) induction of anesthesia, end of surgery, 2 hours and 24 hours after end of surgery
ECG | Screening, 2 hours and 24 hours after end of surgery
  Not mandatory for pediatric patients
Urinalysis | Immediately before or after induction of anesthesia (depending on routine procedures) and 24 hours after surgery
  Not mandatory for pediatric patients
Local and Systemic Tolerance | After each administration of study drug
(Serious) Adverse Events | From signing informed consent until 28 days follow up

CONTACTS AND LOCATIONS:
Overall Officials: Akiyoshi Namiki, MD, PhD, Study Chair — Emeritus Professor Sapporo Medical University; CEO, Otaru City Hospitals, Hokkaido, Japan
Locations (4):
- Japan (4):
  - Sapporo Medical University, School of Medicine, Sapporo, Hokkaido
  - Okayama University, Okayama
  - National Center for Child Health and Development, Tokyo
  - Tokyo Women's Medical University, Tokyo